CLINICAL TRIAL: NCT01117831
Title: An Analysis of Variables That Affect Quality of Diabetes Control in Puerto Rico
Brief Title: An Analysis of Diabetes Control in Puerto Rico
Status: Completed | Type: Observational
Sponsor: Center for Diabetes Control, Inc. (Industry)
Collaborators: Novo Nordisk A/S (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Efrain Rodriguez-Vigil, MD, Medical Director, Center for Diabetes Control, Inc.
Other Study IDs: CD0108
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus; Arterial Hypertension; Hypercholesterolemia
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Epidemiological intervention — An analysis of 600 diabetic patients in the Island of PR to evaluate metabolic control.

SUMMARY:
Project: An analysis of Diabetes Control in Puerto Rico Hypothesis: This project seeks to determine the causes for: i) poor adherence to prescribed treatment by patients, ii) low compliance by providers with national guidelines iii) barriers impose by health insurance in control of diabetes mellitus iv) effectiveness of a disease management program for treatment adherence by patients.

DETAILED DESCRIPTION:
Method (s) The study will consist of three phases:

i) assessment phase,

ii) multimedia health education campaign for patients, providers and local health insurances for adherence improvement

iii) reassessment phase.

Target Population:

Phase I: 600 Hispanic, male and female, residents of Puerto Rico with a diagnosis of type 1 and 2 diabetes mellitus older than 18 of age.

Phase II: 600 patients identified in phase I with individualize health education interventions on the importance of adherence to prescribed medical treatment. 2) Spanish speaking population of Puerto Rico, health service providers, and health insurance companies through a multimedia health education campaign.

Phase III: reassessment of the 600 patients of Phase I.

Data Collection Tools:

i) Demographic information will be obtained by an interview questionnaire. Patients will be assigned a control number automatically by the data system.

ii) Laboratory blood samples for A1C, lipids (total cholesterol, triglycerides and HDL cholesterol), and serum creatinine.

iii) A comprehensive educational adherence program with different media strategies such as: radio spots, newspaper articles, public service announcements, telemedicine services.

Data Analysis: Data will be analyzed using SPSS for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 and 2 diabetic patients older tha 18 years old

Exclusion Criteria:

* 1. Hemophilia.
* 2. Persons younger than 18.
* 3. Persons in research studies of some drug.
* 4. Persons using steroids.
* 5. Patients with acute infections.
* 6. Pregnant diabetic patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This epidemiologic study will analyzed a 600 type 1 and 2 Diabetic patients under medication. The populations to be analyzed is composed of female and male subjects under therapy with anti diabetic medication. The population will be selected from four high density cities in the Island of Puerto Rico. Puerto Ricans are considered as hispanic populations with a mix of white hispanic, african people on a basis of indians ancestry. Subjects will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood sugar control | 2 years
  Numbers of Patients with Hg A1C on control (less than 7%). Those with A1c greater than 7% will be considered as not meeting the goal
Blood pressure control | 2 years
  Blood Pressure Control: Patients will be considered out of blood pressure control if they have a systolic blood pressure greater than 130 mm Hg or a diastolic blood pressure greater than 80 mg Hg
Lipids goal achievement | 2 years
  The following lipids results will be considered out of goal for this population: LDL cholesterol greater than 100 mg/dL, HDL cholestero lower than 40 mg/dL in male and lower than 50 mg/dL in women, and serum triglycerides greater than 150 mg/dL

SECONDARY OUTCOMES:
Achievement of National Clinical Practice Recommendations among Puerto Rican Population with Diabetes Mellitus | 2 years
  Type of therapies used by these populations and their relationship with out of goals outcome.

OTHER OUTCOMES:
Achievement of National Clinical Practice Recommendations among Puerto Rican Population with Diabetes Mellitus | 1 year
  Outcome measure assessment: Descriptive analysis will be computed to describe the demographic and health services characteristic of the participants.
  Bivariate analysis using contingency tables and the Pearson Chi-square test and independent samples t-tests will be conducted to determine whether or not there were differences between adults with diabetes and A1C levels lower than 7% and those with A1C levels greater than 7% in term of demographics, health services characteristics, health insurance type, type of providers, type of medication (insulin or pills) and comorbidities. For statistical analysis, alpha will be set at p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Rodriguez-Vigil, MD, Principal Investigator — Center for Diabetes Control, Inc.

IPD SHARING:
Plan to Share IPD: Yes
National Journal, Physician meeting, Press release
Supporting Information: CSR
Time Frame: 2 years